CLINICAL TRIAL: NCT06718920
Title: Single-center Observational Study to Characterize Adverse Childhood Experiences (ACE) in Patients With Multiple Sclerosis and Their Impact on Quality of Life, Disease Coping Strategies, and Adherence to Disease Course-modifying Therapies
Brief Title: Adverse Childhood Experiences in Patients With MS: Impact on Quality of Life and on Coping Strategies Towards the Disease and Its Treatment
Acronym: ACE-MS
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mirabella Massimiliano, Associate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6791
Record Dates: First submitted 2024-11-21; First posted 2024-12-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: ACE; multiple sclerosis; treatment adherence; adverse childhood experiences; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients referred to the Multiple Sclerosis Center of the Agostino Gemelli IRCCS: Patients diagnosed with multiple sclerosis between 2014 and 2024, referring to the Multiple Sclerosis Center of the Agostino Gemelli IRCCS

SUMMARY:
The goal of this observational study is to evaluate the presence of adverse childhood experiences (ACE) in patients with Multiple Sclerosis. The main questions it aims to answer are:

* Does the presence of ACE impact on quality of life of patients with multiple sclerosis?
* Does it influence how the patients cope with the disease and with disease course-modifying therapies? During follow up visits, planned as part of their regular medical care, participants will answer survey questions on a tablet .

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic inflammatory, demyelinating, and neurodegenerative disease of the central nervous system, typically affecting young adults. Its etiopathogenesis is multifactorial, with the interaction of genetic susceptibility and environmental risk factors. Among these, childhood trauma and other forms of adverse childhood experiences (ACE) such as divorce or parental loss have been called out as possible risk factors in the development of MS and disease relapse.

Adverse Childhood Experiences are a heterogeneous group of negative experiences occurred during childhood, that may have an unfavorable impact on the later course of life in terms of physical and mental health. These effects may be related to changes in the prefrontal, limbic, and hypothalamic-pituitary-adrenal areas and may cause repercussions on the immune system, as documented on experimental models of autoimmune encephalitis. In addition to that, a history of ACE has been associated with the development of poor coping strategies during adulthood . Since multiple sclerosis represents a chronic and progressive disease, the kind of coping strategies developed from childhood may affect how the patient perceives the disease and may affect his or her adherence to treatment.

To date, data on the prevalence of traumatic events during childhood in patients with Multiple Sclerosis are limited to a few studies, while the impact of such events on how the patient copes with the diagnosis of disease and acceptance of therapy. has not yet been explored.

This study represents a preliminary analysis of the impact of ACE in a cohort of multiple sclerosis patients and aims to evaluate how early negative life experiences may affect patients' coping strategies towards the disease and their compliance to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years;
* Diagnosis of relapsing-remitting multiple sclerosis according to McDonald criteria (2017 revisions) made between 2014 and 2024.
* Signature of informed consent

Exclusion Criteria:

* Presence of language barrier
* Presence of conditions that prevent or limit understanding and proper completion of questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 Multiple Sclerosis patients referred to the Multiple Sclerosis Center of the Agostino Gemelli IRCCS University Polyclinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of ACE in a cohort of patients with relapsing-remitting multiple sclerosis | At enrollement
  The patients will answer to questionnaires provided on an electronic tablet during regular follow up neurological visits.
  The presence of adverse childhood experiences will be explored through the completion of a specific questionnaire:
  Childhood Trauma Questionnaire (CTQ): score 0-28 Higher scores mean higher probability to have experienced ACE
To assess the prevalence of ACE in a cohort of patients with relapsing-remitting multiple sclerosis | At enrollement
  The patients will answer to questionnaires provided on an electronic tablet during regular follow up neurological visits.
  The presence of dysfunctional parenting during childhood will be explored through the completion of the Measure of Parental Style (MOPS) questionnaire (score 0-28): higher scores mean higher probability to have experienced dysfunctional parenting, leading to ACE

SECONDARY OUTCOMES:
To correlate the impact of ACE on quality of life and general distress | 1 year
  Quality of life and general distress will be assessed through Brief Symptom Checklist (BSC): score 0-53, higher scores mean higher distress and worse quality of life
To correlate the impact of ACE on how the patient perceives and copes with the disease | 1 year
  Quality of life and physician-patient relationship satisfaction will be assessed through patient reported outcomes
To correlate the impact of ACE on treatment adherence | 1 year
  Treatment satisfaction and compliance will be assessed through patient reported otcomes
To correlate the impact of ACE on disease treatment | 1 year
  To explore treatment satisfaction through the analysis of the number of treatment switches for poor tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corallo F, Bonanno L, Di Cara M, Rifici C, Sessa E, D'Aleo G, Lo Buono V, Venuti G, Bramanti P, Marino S. Therapeutic adherence and coping strategies in patients with multiple sclerosis: An observational study. Medicine (Baltimore). 2019 Jul;98(29):e16532. doi: 10.1097/MD.0000000000016532. PMID 31335734
- [Background] Sheffler JL, Piazza JR, Quinn JM, Sachs-Ericsson NJ, Stanley IH. Adverse childhood experiences and coping strategies: identifying pathways to resiliency in adulthood. Anxiety Stress Coping. 2019 Sep;32(5):594-609. doi: 10.1080/10615806.2019.1638699. Epub 2019 Jul 9. PMID 31288568
- [Background] Nusslock R, Miller GE. Early-Life Adversity and Physical and Emotional Health Across the Lifespan: A Neuroimmune Network Hypothesis. Biol Psychiatry. 2016 Jul 1;80(1):23-32. doi: 10.1016/j.biopsych.2015.05.017. Epub 2015 Jun 4. PMID 26166230
- [Background] Khaw YM, Majid D, Oh S, Kang E, Inoue M. Early-life-trauma triggers interferon-beta resistance and neurodegeneration in a multiple sclerosis model via downregulated beta1-adrenergic signaling. Nat Commun. 2021 Jan 4;12(1):105. doi: 10.1038/s41467-020-20302-0. PMID 33397973
- [Background] McEwen BS. In pursuit of resilience: stress, epigenetics, and brain plasticity. Ann N Y Acad Sci. 2016 Jun;1373(1):56-64. doi: 10.1111/nyas.13020. Epub 2016 Feb 25. PMID 26919273
- [Background] Hepgul N, Pariante CM, Dipasquale S, DiForti M, Taylor H, Marques TR, Morgan C, Dazzan P, Murray RM, Mondelli V. Childhood maltreatment is associated with increased body mass index and increased C-reactive protein levels in first-episode psychosis patients. Psychol Med. 2012 Sep;42(9):1893-901. doi: 10.1017/S0033291711002947. Epub 2012 Jan 20. PMID 22260948
- [Background] Eid K, Bjork MH, Gilhus NE, Torkildsen O. Adverse Childhood Experiences and the Risk of Multiple Sclerosis Development: A Review of Potential Mechanisms. Int J Mol Sci. 2024 Jan 26;25(3):1520. doi: 10.3390/ijms25031520. PMID 38338799
- [Background] Spitzer C, Bouchain M, Winkler LY, Wingenfeld K, Gold SM, Grabe HJ, Barnow S, Otte C, Heesen C. Childhood trauma in multiple sclerosis: a case-control study. Psychosom Med. 2012 Apr;74(3):312-8. doi: 10.1097/PSY.0b013e31824c2013. Epub 2012 Mar 9. PMID 22408134
- [Background] Nikulina V, Widom CS. Child maltreatment and executive functioning in middle adulthood: a prospective examination. Neuropsychology. 2013 Jul;27(4):417-427. doi: 10.1037/a0032811. PMID 23876115